CLINICAL TRIAL: NCT03816462
Title: Reversing the Negative Cardiovascular Effects of Weight (ReNEW) Clinic Cohort Study
Brief Title: ReNEW Clinic Cohort Study
Acronym: ReNEW
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00056175
Record Dates: First submitted 2019-01-22; First posted 2019-01-25 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Hypertension; Prehypertension; Obesity; Overweight; Left Ventricular Hypertrophy; Elevated Blood Pressure
MeSH Terms: conditions — Hypertension; Prehypertension; Obesity; Overweight; Hypertrophy, Left Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an ongoing, prospective cohort study of children and young adults who are evaluated in the Reversing the Negative Effects of Weight on the Heart (ReNEW) Clinic at Johns Hopkins University.

Demographic and clinical data of patients who agree to participate are obtained via chart review and entered into a longitudinal clinic registry.

ELIGIBILITY:
Inclusion criteria:

* Children and young adults with overweight or obesity referred for evaluation of elevated blood pressure in the ReNEW Clinic at Johns Hopkins University are eligible.

Exclusion Criteria:

* Children who are wards of the state or who are non-English speaking without an in-person interpreter accompanying them to the clinic visit.

Max Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children between birth and 22 years of age with overweight or obesity referred for evaluation of elevated blood pressure in the ReNEW Clinic at Johns Hopkins University
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2026-01 (Actual); Study Completion 2026-01 (Actual)

PRIMARY OUTCOMES:
Demographic and clinical data obtained via chart review | 20 years
  This is a clinic based registry of cardiovascular disease risk data from participants to be collected over time.

CONTACTS AND LOCATIONS:
Overall Officials: Tammy M Brady, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Wen W, Psoter KJ, Solomon BS, Urbina EM, Brady TM. Accuracy and Performance of Triage Blood Pressure Measurements in A Real-World Clinic Setting. J Pediatr. 2024 Jun;269:113962. doi: 10.1016/j.jpeds.2024.113962. Epub 2024 Feb 17. PMID 38369238
- [Derived] Ducharme-Smith K, Brady TM, Vizthum D, Caulfield LE, Mueller NT, Rosenstock S, Garcia-Larsen V. Diet quality scores associated with improved cardiometabolic measures among African American adolescents. Pediatr Res. 2022 Sep;92(3):853-861. doi: 10.1038/s41390-021-01893-w. Epub 2021 Dec 16. PMID 34916627
- See also: Please visit the above link for more information. To make an appointment at the ReNEW Clinic, please call 410-955-1247. — https://www.hopkinsmedicine.org/johns-hopkins-childrens-center/what-we-treat/specialties/nephrology/obesity-hypertension-clinic